CLINICAL TRIAL: NCT00280579
Title: Cyanide Poisoning in Fire Victims
Status: Withdrawn | Type: Observational
Why Stopped: Not sufficient time to conduct the study
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: KF 01-277/99
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cases: Cases would have had their blood cyanide concentration measured

SUMMARY:
Aim: To determine the incidence of cyanide poisoning in fire victims.

20 consecutive patients will have the rest of their blood sample analyzed for cyanide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Exposed to smoke from fire and admitted to hospital

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Study Completion 2007-01

PRIMARY OUTCOMES:
Cyanide concentration | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Erik C. Jansen, DMSC, Study Chair — Department of anesthesia, 4231, Center of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Department of Anaesthesia 4231, Centre of Head and Orthopaedics, Copenhagen University Hospital Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Lawson-Smith P, Jansen EC, Hilsted L, Hyldegaard O. Effect of hyperbaric oxygen therapy on whole blood cyanide concentrations in carbon monoxide intoxicated patients from fire accidents. Scand J Trauma Resusc Emerg Med. 2010 Jun 15;18:32. doi: 10.1186/1757-7241-18-32. PMID 20550698